CLINICAL TRIAL: NCT05283096
Title: French Survey on Patients' Practices, Knowledge and Beliefs About Diet in Chronic Inflammatory Rheumatic Diseases (Rheumatoid Arthritis, Psoriatic Arthritis, Spondylarthritis)
Brief Title: Survey About Diet in Chronic Inflammatory Rheumatic Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ALIRIC
Record Dates: First submitted 2022-02-05; First posted 2022-03-16 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-03

CONDITIONS: Rheumatic Disease; Rheumatic Disorder; Inflammatory Rheumatism; Rheumatoid Arthritis; Psoriatic Arthritis; Spondyloarthritis; Spondylitis, Ankylosing; Diet Habit; Feeding Behavior
Keywords: Survey; Questionnaire; Diet; Inflammatory Rheumatism
MeSH Terms: conditions — Rheumatic Diseases; Rheumatic Fever; Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylarthritis; Spondylitis, Ankylosing; Feeding Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic inflammatory rheumatic disease
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire about beliefs on food and diet in rheumatic diseases, and if a diet was tried what effect it had on health and rheumatism

SUMMARY:
A French Survey on patients' practices, knowledge and beliefs about diet in chronic inflammatory rheumatic diseases (rheumatoid arthritis, psoriatic arthritis, spondylarthritis) Use of a questionnaire about what patients have heard concerning diet and rheumatism, what kind of diet they tried eventually and how it affected their health and disease

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with chronic inflammatory rheumatism (rheumatoid arthritis, spondylarthritis, psoriatic arthritis) according to the diagnostic criteria commonly admitted
* Patient followed in the rheumatology department of the University Hospital of Poitiers (France)
* Free patient, without guardianship or tutelage or subordination
* Patient not opposing to participate in the study

Exclusion Criteria:

* Patient withdrawing consent
* Patient who does not meet criteria for chronic inflammatory disease (rheumatoid arthritis, spondylarthritis, psoriatic arthritis) according to the diagnostic criteria commonly admitted after examination of medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed in the rheumatology department of the University Hospital of Poitiers (France) for chronic inflammatory rheumatism, going for consultation or hospitalisation for usual care
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence (rate) of patients with chronic inflammatory rheumatism who have changed their dietary practices since being diagnosed. | 6 months
  To assess the prevalence of dietary changes in patients with chronic inflammatory rheumatism (rheumatoid arthritis, spondylarthritis and psoriatic arthritis) using a questionnaire

SECONDARY OUTCOMES:
Rate of patients believing that diet affects their rheumatism | 6 months
  To describe the practices, knowledge and beliefs about diets of patients with chronic inflammatory rheumatism using a questionnaire
Rate of patients following each specific diet (gluten free, vegetarian, dairy products free, ...) | 6 months
  To describe the practices, knowledge and beliefs about diets of patients with chronic inflammatory rheumatism using a questionnaire
Comparison of the rates of patients believing that diet affects their rheumatism, between each subgroup of rheumatism | 6 months
  To compare dietary beliefs, knowledge and practices between different patient subgroups (rheumatoid arthritis, spondyloarthritis, psoriatic arthritis) with their answers to the questionnaire
Comparison of the rates of patients following each specific diet (gluten free, vegetarian, dairy products free, ...) between each subgroup of rheumatism | 6 months
  To compare dietary beliefs, knowledge and practices between different patient subgroups (rheumatoid arthritis, spondyloarthritis, psoriatic arthritis) with their answers to the questionnaire
Comparison of the rates of patients who were able to stop a part of their treatment between the diet and non-diet groups | 6 months
  To compare drug management and disease activity between different dietary practices (with and without practice modification) with their answers to the questionnaire
Comparison of disease activity by the level of C reactive protein, DAS 28, ASDAS and BASDAI between the diet and non-diet groups | 6 months
  To compare drug management and disease activity between different dietary practices (with and without practice modification) with their answers to the questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, Nouvelle-Aquitaine, France

IPD SHARING:
Plan to Share IPD: Undecided